CLINICAL TRIAL: NCT00377715
Title: Phase 2, Double-Blind, Placebo-Controlled Study of Oral Dimebon in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Double-blind, Placebo-controlled Study of Oral Dimebon in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIM02
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer's Disease
Keywords: Dimebon, Alzheimer's Disease, Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog)
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dimebon (Experimental): Dimebon 20 mg three times a day x 26 weeks
  Interventions: Drug: Dimebon
- Placebo (Placebo Comparator): Placebo 20 mg three times a day x 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimebon
  Arms: Dimebon
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and potential benefit of Dimebon as compared to placebo in patients with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females greater than or equal to 50 years of age.
2. Diagnosis of Alzheimer's Disease according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV TR) and Mini Mental State Exam between 10 and 24, inclusive and Modified Hachinski Ischemia Score less than or equal to 4.
3. Brain imaging such as MRI and/or CT within one year of enrollment.
4. Subjects must have a guardian or caregiver who assists the subject at least 5 days per week (at least 3 hours/day).
5. Subjects must be able to cooperate with drug administration (including the ability to ingest oral medications) and study procedures and abide by study restrictions.
6. Subjects must have at least 6 years of prior education and should have previously (in pre-Alzheimer's condition) been capable of reading, writing and communicating effectively with others.
7. Subjects must be willing and able to give informed consent or have a mentally competent legal representative authorized to provide informed consent on their behalf.
8. Residence in an assisted care facility is allowed if subject is living independently.

Exclusion Criteria:

1. Major structural brain disease
2. Major medical illness or unstable medical condition within 6 months of screening that may interfere with the subject's ability to comply with study procedures and abide by study restrictions.
3. Residence in a nursing home or assisted care facility that provides the subject with 24-hour care and supervision.
4. Women who are pregnant, nursing, or if of child-bearing potential not using a medically accepted, highly effective method of birth control.
5. Active alcohol dependence or drug abuse.
6. Use of the following medications within 60 days prior to enrollment:cognition enhancing agents, narcotic analgesics, low potency neuroleptics, antihypertensive agents with frequent Central Nervous System (CNS) side effects, anti-Parkinsonian medications, medications with central anticholinergic activity, medications for epilepsy, lithium.
7. Participation in an investigational drug or device study within 30 days prior to study entry, or 60 days prior to study entry if the investigational drug study involved therapy for Alzheimer's Disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-09; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - cognitive subscale | 26 weeks

SECONDARY OUTCOMES:
Clinical Global Impression of Change | 26 weeks
Safety Assessed By Number of Participants With Adverse Events | 26 weeks
  Adverse events will be assessed through physical examinations, electrocardiograms, and clinical laboratory data (chemistry panel, complete blood count (CBC) with differential, and urinalysis). The incidence of adverse events will be summarized by severity and relationship to study treatment.
Pharmacokinetic (PK) parameter of Dimebon: Cmax | Week 1, 2, 6, 12, 18, 24. Blood PK samples will be obtained pre-dose and 1 hour post-dose for each timepoint.
  Cmax: Maximum concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Research Center of Russian Academy of Medical Sciences, Moscow, Moscow, Russia

REFERENCES:
- [Derived] Doody RS, Gavrilova SI, Sano M, Thomas RG, Aisen PS, Bachurin SO, Seely L, Hung D; dimebon investigators. Effect of dimebon on cognition, activities of daily living, behaviour, and global function in patients with mild-to-moderate Alzheimer's disease: a randomised, double-blind, placebo-controlled study. Lancet. 2008 Jul 19;372(9634):207-15. doi: 10.1016/S0140-6736(08)61074-0. PMID 18640457